CLINICAL TRIAL: NCT06417554
Title: A Phase IB /II, Multicenter, Open-Label Study of Safety, Tolerability and Efficacy of SHR-A2102 for Injection With or Without Antitumor Therapy in Subjects With Advanced Solid Tumors
Brief Title: A Trial of SHR-A2102 With or Without Antitumor Therapy in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A2102-201
Record Dates: First submitted 2024-04-26; First posted 2024-05-16 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A: SHR-A2102 + Adebrelimab injection (Experimental)
  Interventions: Drug: SHR-A2102 ; Adebrelimab injection
- Treatment group B: SHR-A2102 (Experimental)
  Interventions: Drug: SHR-A2102

INTERVENTIONS:
Drug: SHR-A2102 — SHR-A2102
  Arms: Treatment group B: SHR-A2102
Drug: SHR-A2102 ; Adebrelimab injection — SHR-A2102 + Adebrelimab injection
  Arms: Treatment group A: SHR-A2102 + Adebrelimab injection

SUMMARY:
The study is being conducted to evaluate the safety, tolerability and efficacy of SHR-A2102 for injection with or without Antitumor Therapy in Advanced Solid Tumors. To explore the reasonable dosage of SHR-A2102 for Advanced Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to give informed consent, have signed informed and able to comply with the treatment plan to visit the tests and other procedural requirements；
2. The age of signing the informed consent is above 18 years old, regardless of gender；
3. The ECOG score is 0 or 1；
4. Expected survival ≥12 weeks
5. Subjects with pathologically confirmed locally advanced unresectable or metastatic solid tumors, stage Ib subjects who have failed standard treatment; Stage II subjects with pathologically confirmed locally advanced unresectable or metastatic solid tumors without systemic antitumor therapy；
6. Provide archived or fresh tumor tissue；
7. At least one measurable lesion according to RECIST v1.1 criteria；
8. Good level of organ function；
9. Male subjects whose partners are women of childbearing age and female subjects who are fertile are required to use highly effective contraceptive methods

Exclusion Criteria:

1. Inadequately treated central nervous system metastases or the presence of uncontrolled or symptomatic active central nervous system metastases；
2. Have previously received antiboy-coupled drugs containing topoisomerase I inhibitors; Stage II was previously treated with PD-1/PD-L1 inhibitors；
3. Systemic antitumor therapy was received 4 weeks before the start of the study；
4. Palliative radiotherapy was completed within 14 days before the first dose; Chest radiotherapy >30 Gy within 6 months prior to initial administration；
5. Toxicity and/or complications of previous antitumor therapy did not return to NCI-CTCAE level ≤1 or exclusion criteria；
6. Systemic immunosuppressive therapy was administered within 14 days prior to the first study；
7. Subjects with known or suspected interstitial pneumonia；
8. ≥ grade 3 immune-related adverse events occurred during previous treatment with immune checkpoint inhibitors；
9. The presence of any active, known, or suspected autoimmune disease；
10. Moderate or severe ascites with clinical symptoms, uncontrolled or moderate or above pleural effusion and pericardial effusion；
11. The presence of clinical cardiac symptoms or diseases that are not well controlled；
12. Any other malignancy diagnosed within the previous 5 years；
13. Subjects who had a severe infection within 28 days prior to the first dose；
14. Active hepatitis B or active hepatitis C；
15. Patients with active tuberculosis infection within 1 year prior to enrollment, or with a history of active tuberculosis infection more than 1 year prior but without formal treatment；
16. History of immune deficiency；
17. Live attenuated vaccines were used within 28 days prior to initial study administration or during the expected study period；
18. Participants who are participating in another clinical study or whose first dose is less than 4 weeks from the end of the previous clinical study (last dose), or five half-lives of the investigational drug, whichever is shorter；
19. Have undergone major surgery other than diagnosis or biopsy within 28 days prior to initial dosing; Minor traumatic surgery within 7 days prior to first dosing; Presence of non-healing wounds or untreated fractures；
20. Severe allergic reactions are known to occur in individuals allergic to any component of SHR-A2102, SHR-1316, or other monoclonal antibody/fusion protein drugs；
21. Female subjects who are pregnant or plan to become pregnant during the study period；
22. The presence of uncontrolled mental illness and other conditions known to affect the completion of the study process, such as alcohol, drug or substance abuse, and criminal detention；
23. In the investigator's judgment, there are any other circumstances that may increase the risk of participating in the study, interfere with the study results, or make participation in the study inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
RP2D | through phase IB completion, an average of 1 years
Incidence and severity of AE； | from Day1 to 90 days after last dose
ORR | 18 months after the last subject was enrolled in the group

SECONDARY OUTCOMES:
DCR(Investigator evaluation) | 18 months after the last subject was enrolled in the group
DoR(Investigator evaluation) | 18 months after the last subject was enrolled in the group
PFS(Investigator evaluation) | 18 months after the last subject was enrolled in the group
OS(Investigator evaluation) | 18 months after the last subject was enrolled in the group
SHR-A2102 and free toxin PK | through study completion, an average of 2 years
SHR-1316 PK | through study completion, an average of 2 years
SHR-A2102 Immunogenicity | through study completion, an average of 2 years
SHR 1316 Immunogenicity | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided